CLINICAL TRIAL: NCT00992329
Title: Impact of Formulation on Ciprofloxacin Oral Absorption
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, James E Polli, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HP-00043432; HHSF223200810030C (Other Grant/Funding Number: DHHS)
Record Dates: First submitted 2009-10-02; First posted 2009-10-09 (Estimated); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Healthy
Keywords: ciprofloxacin; pharmacokinetics; formulation
MeSH Terms: interventions — Ciprofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- ciprofloxacin tab1 (Experimental): formulation 1
  Interventions: Drug: ciprofloxacin
- ciprofloxacin tab2 (Experimental): formulation 2
  Interventions: Drug: ciprofloxacin
- ciprofloxacin tab 3 (Experimental): formulation 3
  Interventions: Drug: ciprofloxacin
- ciprofloxacin reference (Active Comparator): reference product
  Interventions: Drug: ciprofloxacin

INTERVENTIONS:
Drug: ciprofloxacin — ciprofloxacin 200mg tablet (single dose)

SUMMARY:
The purpose of this research is to see if certain tablet formulation factors affect oral drug absorption. Medications taken by mouth, such as tablets, need to be absorbed into the body in order to do any good. Tablets contain a drug, but also contain non-drug ingredients that are called excipients or fillers. Excipients in the tablet, and the way in which the tablet is manufactured, both can impact how much drug is absorbed into the body. That is, tablet formulation factors can cause a tablet to be effective or not effective.

Tablets in this research contain the drug ciprofloxacin hydrochloride. Ciprofloxacin is an antibiotic to treat infections, such as lung infections. This drug is being used since it has low water solubility and is probably sensitive to tablet formulation factors.

DETAILED DESCRIPTION:
Dogs and humans exhibit differences in gastrointestinal physiology. The development of pharmaceuticals for both humans and dogs typically depends upon pharmacokinetic studies in the other species. Product design and quality attributes for dogs (and for humans)generally conduct such extrapolations in a simplistic fashion, without a systematic account of the differential intestinal physiology between dog and human. This project aims to elucidate product quality differences between human and dog oral solid dosage forms as a result of the differential physiology between the two specifies. This insight will facilitate the regulation of canine medicines by highlighting how product standards for human medicines are either too liberal or too restrictive for canine medicines.

Ciprofloxacin hydrochloride will be used as a model poorly soluble drug. A range of immediate-release (IR) tablets will be formulated to map the design space. Formulations will be fast, medium, and slow, with respect to dissolution rate of drug. Ciprofloxacin is expected to exhibit formulation-dependent pharmacokinetics, which is additionally impacted by the differential physiology between dog and humans. In particular, the investigators anticipate a greater sensitivity to formulation for dogs than for humans. Consequently, the investigators anticipate dogs to be more sensitive to formulations, where such critical formulation factors must be considered in canine product design and regulation.

Objectives: 1) The primary objective of this human study is to assess whether specific formulation factors impact the rate and extent of ciprofloxacin oral absorption, as well as the absolute absorption profile of ciprofloxacin. 2) The secondary objective is to assess if dogs exhibit a greater sensitivity to formulation than do humans.

Hypotheses: The investigators anticipate that humans exhibit a modest sensitivity to specific tablet formulation factors. 1) Hence, the hypothesis of this human study is that humans do not exhibit a sensitivity to specific formulation factors and show no in vitro - in vivo correlation to dissolution rate. 2) Alternative hypothesis is that humans do exhibit a sensitivity to specific formulation factors and show an in vitro - in vivo correlation to dissolution rate.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age 18-55
* Healthy volunteers: Subjects in good health, as determined by screening evaluation that is not greater than 30 days before the first drug study visit
* Willing to avoid caffeine containing products 24 hours prior to and day of study visits
* Willing to stop all OTC medications for 24 hours prior to and during study visits
* Able to provide informed consent

Exclusion Criteria:

* Presence of significant medical disease (including cardiovascular, pulmonary, hematologic, endocrine, immunologic, neurologic, gastrointestinal or psychiatric)
* Presence of hepatic, renal disease
* Pregnant women, breast feeding or trying to become pregnant
* Excessive alcohol use (i.e. current physical, behavioral, or personal manifestations related to the abuse or dependency on alcohol)
* Routine use (i.e. daily or weekly) prescription medication except birth control pills
* Routine use (i.e. daily or weekly) use of acid blockers, antacids, anti-diarrhea, stimulants, appetite suppressants, or anti nausea medication or other drugs that modulate GI function
* Currently taking ciprofloxacin or tizanidine
* Allergic to ciprofloxacin or any quinolone-type antibiotic (e.g. levofloxacin)
* Currently taking a corticosteroid drug (e.g. prednisone)
* Had a kidney, heart, or lung transplant
* Any condition in which in the opinion of the PI or medical physician would increase risk to the subject or interfere with the integrity of the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2013-01; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Amount of ciprofloxacin absorbed | 10 hours
  Blood samples will be collected to measure level of ciprofloxacin.

SECONDARY OUTCOMES:
Difference between humans and dogs in the amount of cipro absorbed. | 10 hours
  Blood samples will be collected to measure level of ciprofloxacin.

CONTACTS AND LOCATIONS:
Overall Officials: James Polli, Principal Investigator — University of Maryland, College Park
Locations (1):
- University of Maryland, Baltimore, Maryland, United States

REFERENCES:
- [Background] Polli JE, Rekhi GS, Augsburger LL, Shah VP. Methods to compare dissolution profiles and a rationale for wide dissolution specifications for metoprolol tartrate tablets. J Pharm Sci. 1997 Jun;86(6):690-700. doi: 10.1021/js960473x. PMID 9188051